CLINICAL TRIAL: NCT05969119
Title: Addition of Pyridostigmine to Conventional Management of Postdural Puncture Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, riham fathy galal, Lecturer of Anesthesia intensive care and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUEZ Med-IRB 1/2023
Record Dates: First submitted 2023-06-28; First posted 2023-08-01 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Postdural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Pyridostigmine Bromide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pyridostigmine (Experimental): Parturients with postoperative PDPH and a VAS score of ≥5 will receive either 60 mg oral Pyridostigmine every 6 hours.
  Interventions: Drug: Pyridostigmine
- Placebo (Placebo Comparator): Parturients with postoperative PDPH and a VAS score of ≥5 will receive placebo tablets similar in shape to pyridostigmine tablets every 6 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyridostigmine — Parturients with postoperative Postdural puncture headache and a Visual analogue scale (VAS score) of ≥5 will receive either 60 mg oral Pyridostigmine every 6 hours or Placebo tablets similar in shape to pyridostigmine tablets every 6 hours.
  Arms: Pyridostigmine
Drug: Placebo — Parturients with postoperative Postdural puncture headache and a Visual analogue scale (VAS score) of ≥5 will receive Placebo tablets similar in shape to pyridostigmine tablets every 6 hours.
  Arms: Placebo

SUMMARY:
Postdural puncture headache (PDPH) is a major complication of neuraxial anesthesia that can occur following spinal anesthesia and with inadvertent Dural puncture during epidural anesthesia. The presence of Pyridostigmine in CSF would be expected to increase the level of acetylcholine in CSF and subsequently in the brain through inhibition of cholinesterase. The increased level of acetylcholine would produce cerebral vasoconstriction.

ELIGIBILITY:
Inclusion Criteria:

* Patients American Society of anesthesiologists' physical status (ASA) II because of pregnancy.
* Patients diagnosed with Postdural puncture headache following intrathecal spinal anesthesia for elective caesarean delivery.

Exclusion Criteria:

1. Patients with PDPH and a visual analog scale (VAS) score <5.
2. Patients with history of chronic headache, cluster headache, migraine, convulsions.
3. Patients with history of cerebrovascular accident, previous neurological diseases.
4. Patients with preeclampsia, eclampsia, coagulopathy.
5. Patients with severe bleeding (>20% of blood volume).
6. Patients undergoing treatment with vasopressors.
7. Patients with bronchial asthma.
8. Patients with arrhythmia, and any type of heart block.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to determine the difference in VAS score between the Pyridostigmine group and the control group. | 15 minutes after sitting upright
  Participants will be asked to report the severity of their headache after sitting upright for 15 minutes, using a 10-cm VAS( Visual analogue scale) where 10 refers to the worst pain at 0 hours.
The primary outcome is to determine the difference in VAS score between the Pyridostigmine group and the control group. | 6 hours
  Participants will be asked to report the severity of their headache after sitting upright for 15 minutes, using a 10-cm VAS( Visual analogue scale) after 6 hours.
The primary outcome is to determine the difference in VAS score between the Pyridostigmine group and the control group. | 12 hours
  Participants will be asked to report the severity of their headache after sitting upright for 15 minutes, using a 10-cm VAS( Visual analogue scale) after 12 hours.
The primary outcome is to determine the difference in VAS score between the Pyridostigmine group and the control group. | 24 hours
  Participants will be asked to report the severity of their headache after sitting upright for 15 minutes, using a 10-cm VAS( Visual analogue scale) after 24 hours.
The primary outcome is to determine the difference in VAS score between the Pyridostigmine group and the control group. | 36 hours
  Participants will be asked to report the severity of their headache after sitting upright for 15 minutes, using a 10-cm VAS( Visual analogue scale) after 36 hours.
The primary outcome is to determine the difference in VAS score between the Pyridostigmine group and the control group. | 48 hours
  Participants will be asked to report the severity of their headache after sitting upright for 15 minutes, using a 10-cm VAS( Visual analogue scale) after 48 hours.
The primary outcome is to determine the difference in VAS score between the Pyridostigmine group and the control group. | 72 hours
  Participants will be asked to report the severity of their headache after sitting upright for 15 minutes, using a 10-cm VAS( Visual analogue scale) after 72hours.

SECONDARY OUTCOMES:
The need for an Epidural blood patch in the Pyridostigmine and control groups. | 72 hours
  An EBP will be performed during the study if the VAS(Visual analogue scale) will be ≥5 after 72 hours from intervention start following parturient approval and consent, or if requested by the parturient at any time during the study.
Appearance of neck stiffness in the Pyridostigmine and control groups. | Before giving the Pyridostigmine or the Placebo
  Appearance of neck stiffness in the Pyridostigmine and control groups and will be recorded after asking the patients by yes or no.
Appearance of neck stiffness in the Pyridostigmine and control groups. | 6 hours after the intervention
  Appearance of neck stiffness in the Pyridostigmine and control groups and will be recorded after asking the patients by yes or no.
Appearance of neck stiffness in the Pyridostigmine and control groups. | 12 hours after the intervention
  Appearance of neck stiffness in the Pyridostigmine and control groups that will be recorded after asking the patients by yes or no.
Appearance of neck stiffness in the Pyridostigmine and control groups. | 24 hours after the intervention
  Appearance of neck stiffness in the Pyridostigmine and control groups and will be recorded after asking the patients by yes or no.
Appearance of neck stiffness in the Pyridostigmine and control groups. | 36 hours after the intervention
  Appearance of neck stiffness in the Pyridostigmine and control groups and will be recorded after asking the patients by yes or no.
Appearance of neck stiffness in the Pyridostigmine and control groups. | 48 hours after the intervention
  Appearance of neck stiffness in the Pyridostigmine and control groups and will be recorded after asking the patients by yes or no.
Appearance of neck stiffness in the Pyridostigmine and control groups. | 72 hours after the intervention
  Appearance of neck stiffness in the Pyridostigmine and control groups and will be recorded after asking the patients by yes or no.
Appearance of Nausea and vomiting in the Pyridostigmine and control groups. | Before giving the Pyridostigmine or the Placebo
  Appearance of Nausea and vomiting in the Pyridostigmine and control groups that will be recorded after asking the patients by yes or no.
Appearance of Nausea and vomiting in the Pyridostigmine and control groups. | 6 hours after the intervention
  Appearance of Nausea and vomiting in the Pyridostigmine and control groups that will be recorded after asking the patients by yes or no.
Appearance of Nausea and vomiting in the Pyridostigmine and control groups. | 12 hours after the intervention
  Appearance of Nausea and vomiting in the Pyridostigmine and control groups that will be recorded after asking the patients by yes or no.
Appearance of Nausea and vomiting in the Pyridostigmine and control groups. | 24 hours after the intervention
  Appearance of Nausea and vomiting in the Pyridostigmine and control groups that will be recorded after asking the patients by yes or no.
Appearance of Nausea and vomiting in the Pyridostigmine and control groups. | 36 hours after the intervention
  Appearance of Nausea and vomiting in the Pyridostigmine and control groups that will be recorded after asking the patients by yes or no.
Appearance of Nausea and vomiting in the Pyridostigmine and control groups. | 48 hours after the intervention
  Appearance of Nausea and vomiting in the Pyridostigmine and control groups that will be recorded after asking the patients by yes or no.
Appearance of Nausea and vomiting in the Pyridostigmine and control groups. | 72 hours after the intervention
  Appearance of Nausea and vomiting in the Pyridostigmine and control groups that will be recorded after asking the patients by yes or no.

CONTACTS AND LOCATIONS:
Locations (1):
- Suez General Hospital, Suez, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
according to the researchers plan